CLINICAL TRIAL: NCT00642720
Title: The Effects of Weekly Administration of 40 mg Pegvisomant or Placebo on Quality of Life and Insulin Sensitivity in Acromegalic Patients With Normal IGF-I Concentrations During Long-Term Treatment With Long-Acting Somatostatin Analogs
Brief Title: Change in Quality of Life After Addition of Weekly 40 mg Pegvisomant/Placebo in Controlled Acromegalic Patients
Acronym: mec-2005-290
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Aart-Jan van der Lely, Erasmus Medical center
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: *P05.1649L; *P05.1649L CCMO
Record Dates: First submitted 2008-03-21; First posted 2008-03-25 (Estimated); Last update posted 2008-03-25 (Estimated); Status verified 2008-03

CONDITIONS: Quality of Life; Acromegaly
MeSH Terms: conditions — Acromegaly | interventions — pegvisomant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- pegvisomant-placebo (Other): patients in this arm received(as addition)for the first 8 weeks Pegvisomant and the later for 8 weeks Placebo. This was divided by a 4 weeks wash-out period.
  Interventions: Drug: Pegvisomant
- placebo-pegvisomant (Other): Patient received for the first 8 weeks Pegvisomant and after a wash out period of 4 weeks the received 8 of placebo treatment
  Interventions: Drug: Pegvisomant

INTERVENTIONS:
Drug: Pegvisomant — if the addition of 40 mg pegvisomant weekly will improve the quality of life of acromegaly patients compared to placebo weekly

SUMMARY:
Study Synopsis Study Title: Double blind, single centre, cross-over study on the effects of weekly subcutaneous administration of 40 mg pegvisomant or placebo on quality of life and insulin sensitivity in acromegalic patients with normal serum IGF-I concentrations during long-term treatment with long-acting somatostatin analogs

Study Objectives:

1. To determine whether the addition of weekly pegvisomant administrations improves quality of life
2. To determine whether the addition of weekly pegvisomant administrations improves insulin sensitivity

Study Population: Acromegalic patients, who have normalized their serum IGF-I levels down to the upper 25 centiles of normality during long-term treatment with monthly injections of a long-acting somatostatin analogue Number of Subjects: 20

Procedures:

* Patients on treatment with Sandostatin LAR (SL) 20 - 30 mg per months i.m. or patients on treatment with Lanreotide autosolution (LA) 90 - 120 mg deep s.c. will be enrolled.
* For 4 months, all subjects will also receive weekly s.c. injections of either placebo or a fixed dose of 40 mg pegvisomant
* After a 4 weeks wash-out period, patients will switch from either placebo to pegvisomant or from pegvisomant to placebo
* Before, and after 2 and 4 months of each treatment period, serum efficacy parameters and quality of life (AcroQol ™/ PASQ™) will be assessed.
* Before and after 4 months of each treatment period, pituitary tumor size and insulin sensitivity (HOMA/SIGMA model) will be assessed. Duration of study: 9 months

Hypothesis:

•We postulate that co-administration of the growth hormone receptor antagonist pegvisomant will improve QoL and insulin sensitivity

DETAILED DESCRIPTION:
Introduction Both lanreotide (Somatulin Autosolution ™ (SL)) and octreotide (Sandostatin LAR ™ (LAR)) are equally effective in controlling disease activity in acromegalic subjects with a normalization of serum insulin-like growth factor-I (IGF-I) levels in roughly 65%. However, SL is injected as a deep intramuscular injection, while LA is injected as a deep subcutaneous injection. Physicians, involved in the treatment of acromegalic patients know that biochemical control of the disease in their patients not necessarily means that all those patients stop complaining. To address these issues, Sonino and co-workers studied with several symptom questionnaires the effects on quality of life (QoL) of SL. Together with a significant decrease in growth hormone (GH) and IGF-I, treatment with SL significantly improved psychological distress, well-being and social fears (1). In another study on the efficacy of the novel GH receptor antagonist pegvisomant to lower serum IGF-I concentrations a questionnaire evaluating five clinical signs and symptoms of acromegaly showed dose dependent significant differences from placebo (2). Recently, Webb and co-workers reported the successful development of a disease-specific questionnaire suitable to measure health-related quality of life in acromegaly (ACROQOL) (3).

No clear biochemical parameter appears to be available that correlates well with disease activity related quality of life (4). At the same time, serum GH concentrations and serum total IGF-I levels, but not QoL, are used as parameters to determine dosing of Sandostatin LAR, or any of the available medical therapies for acromegaly (5-8).

The growth hormone receptor antagonist pegvisomant as monotherapy once daily normalizes IGF-I in virtually all acromegalics (9;10), but pegvisomant monotherapy is also very costly. Recently, we reported the results of a 42-week dose-finding study on the efficacy of the combination of long-acting somatostatin analogues once monthly and pegvisomant once weekly in 26 patients with active acromegaly. Pegvisomant dose was increased until IGF-I levels normalized or until a weekly dose of 80 mg was reached. IGF-I levels normalized in 25 (95 %) with a median weekly dose of 60 mg pegvisomant. There were no signs of pituitary tumor growth but mild elevations in liver enzymes were observed in 10 patients (38%) (11). One of the potential advantages of combining pegvisomant with somatostatin analogues is that pegvisomant monotherapy improves insulin sensitivity compared to somatostatin analogues (12;13), although it is unclear yet whether or not long-term pegvisomant administration would improve insulin sensitivity in normal subjects (13;14). Therefore, one might expect that pegvisomant monotherapy has beneficial effects on insulin sensitivity, compared to the combination of both pegvisomant and somatostatin analogues, as the latter ones decrease insulin sensitivity by several mechanisms (13;15).

Conclusion:

* So-called biochemically well controlled acromegalic subjects with normal serum IGF-I concentrations frequently still have an impaired QoL.
* These subjects, when controlled by long-acting somatostatin analogs have impaired insulin sensitivity because of the pharmacological properties of these somatostatin analogs.
* We postulate that co-administration of the growth hormone receptor antagonist pegvisomant will improve QoL and insulin sensitivity

Objectives:

1. To determine whether the addition of weekly pegvisomant administrations improves quality of life
2. To determine whether the addition of weekly pegvisomant administrations improves insulin sensitivity

Description of procedures:

* Patients on treatment with Sandostatin LAR (SL) 20 - 30 mg per months i.m. or patients treated with Lanreotide autosolution (LA) 90 - 120 mg deep s.c. will be enrolled.
* For 4 months, and after randomization, all subjects will also receive weekly s.c. injections of either placebo or a fixed dose of 40 mg pegvisomant
* After a 4 weeks wash-out period, patients will switch from either placebo to pegvisomant or from pegvisomant to placebo
* Before, and after 2 and 4 months of each treatment period, serum efficacy parameters and quality of life (AcroQol ™ , general QoL questionaire and PASQ Signs and Symptoms) will be assessed.
* Before and after 4 months of each treatment period, pituitary tumor size and insulin sensitivity (HOMA/SIGMA model (16)) will be assessed.

Subjects Twenty acromegalic subjects who are seen at regular intervals at our out-patient facilities will be asked to participate. All subjects will be seen at the Clinical Research Unit.

Inclusion criteria:

* Active acromegaly.
* Serum total IGF-I levels must have been normalized during long-term treatment with long-acting somatostatin analogs
* Age between 18 and 80

Exclusion criteria:

* Any contra-indication for the use of long-acting somatostatin analogs, as e.g. the use of anti-coagulants.
* Subjects with pituitary tumors that compress the optic chiasm
* Patients with insulin dependent diabetes
* Patients with cancer
* Patients with kidney- or liver function disturbances
* Fertile female patients that refuse to take contraceptives during the study

Study procedures Visit 1; baseline (week 0; 1 day prior to next monthly injection of long-acting SRIF analog))

* Review inclusion and exclusion criteria
* Obtain written informed consent
* Conduct a medical history and physical examination; record vital signs.
* Blood sampling: fasting IGF-I, insulin, GH, glucose, HbA1c, liver functions, lipid profile, free fatty acids, pegvisomant levels, pregnancy test in females.
* QoL assessment (AcroQol™/PASQ ™)
* MRI (recent MRI of < 3 months is also acceptable)
* Injection of the usual SL or LA dose
* randomization
* Start of weekly injections of 40 mg pegvisomant or placebo (16 injections in total)

Visit 2, 3 (week 8 and 16; one day prior of weekly study drug/placebo injection)

* Blood sampling: fasting IGF-I, insulin, GH, glucose, HbA1c, liver functions, lipid profile, free fatty acids, pegvisomant levels
* QoL assessment (AcroQol™/PASQ ™)
* After week 16, all patients have their 4 weeks wash-out period
* MRI

Visit 4 (week 20; end of wash-out)

* Blood sampling: fasting IGF-I, insulin, GH, glucose, HbA1c, liver functions, lipid profile, free fatty acids, pegvisomant levels
* Return of study medication for drug accountability
* QoL assessment (AcroQol™/PASQ ™)
* Start of second co-treatment period with weekly s.c injections of either placebo or 40 mg fixed-dose pegvisomant (16 weekly injections)

Visit 5, 6 (week 28 and 36; one day prior of weekly study drug/placebo injection)

* Blood sampling: fasting IGF-I, insulin, GH, glucose, HbA1c, liver functions, lipid profile, free fatty acids, pegvisomant levels
* Return of study medication for drug accountability
* QoL assessment (AcroQol™/PASQ ™)
* MRI

ELIGIBILITY:
Inclusion Criteria:

* Active acromegaly.
* Serum total IGF-I levels must have been normalized during long-term treatment with long-acting somatostatin analogs
* Age between 18 and 80

Exclusion Criteria:

* Any contra-indication for the use of long-acting somatostatin analogs, as e.g. the use of anti-coagulants.
* Subjects with pituitary tumors that compress the optic chiasm
* Patients with insulin dependent diabetes
* Patients with cancer
* Patients with kidney- or liver function disturbances
* Fertile female patients that refuse to take contraceptives during the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2006-10; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
To assess if the addition of pegvisomant weekly will improve Quality of life (QoL). QoL will be assessed by the PASQ and AcroQol questionnaires | at 8 and 16 weeks of treatment

SECONDARY OUTCOMES:
If the addition of pegvisomant will improve metabolic parameters such as Insulin sensitivity, lipids, Glucose, IGF-I ect. | at 8 and 16 weeks